CLINICAL TRIAL: NCT05153460
Title: Pilot Clinical Evaluation of Dozee VS in Hospital Patients
Brief Title: Pilot Clinical Evaluation of Dozee VS, a Contactless Continuous Vital Parameters Monitoring System in Hospital Patients
Acronym: DZUSFDA21
Status: Terminated | Type: Observational
Why Stopped: Site unable to recruit subjects
Sponsor: Turtle Shell Technologies Pvt. Ltd. (Industry)
Collaborators: Louisiana State University Health Sciences Center in New Orleans (Other); HealthMinds (Unknown)
Responsible Party: Sponsor
Other Study IDs: DozeeUSFDA2021; STUDY00001760 (Other: Louisiana State University Health Sciences Center)
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: No Specific Medical Conditions or Disease States
Keywords: Continuous Monitoring, Ballistocardiography, HR, RR, DozeeVS
MeSH Terms: interventions — Telemetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Single Arm Study (Cohort): All participants will be on standard telemetry monitoring for Heart Rate and Respiration Rate using the gold standard (Electrocardiography and Capnography respectively).
  In addition, two contactless monitoring devices will be placed on the patient bed to measure data simulataneously. These devices include EarlySense (USFDA approved ballistocardiography device) and Dozee VS (Investigational Device).
  Interventions: Device: Telemetry and manual monitoring vs Contactless monitoring devices

INTERVENTIONS:
Device: Telemetry and manual monitoring vs Contactless monitoring devices — All participants will be on standard telemetry monitoring for Heart Rate, Respiration Rate and movements using the gold standard (Electrocardiography and Capnography respectively).
  In addition, two contactless monitoring devices will be placed on the patient bed to measure data simultaneously. These devices include EarlySense (USFDA approved ballistocardiography device) and Dozee VS (Investigational Device).
  Other Names: EarlySense; Dozee VS

SUMMARY:
The Dozee VS device developed by Turtle Shell Technologies Pvt. Ltd., is a contactless continuous vital parameters monitoring system. It is designed for continuous and contactless measurement of Heart Rate (HR) and Respiratory Rate (RR). The device uses the concept of ballistocardiography and deploys piezoelectric sensors to capture the micro-vibrations originating from cardiac contractions, upper respiratory tract activity and body movements. This data is then analyzed by a proprietary algorithm and the values of the vital parameters - Heart Rate (HR) and Respiratory Rate (RR) are generated. The captured vital parameters can be accessed remotely via a dashboard which can be accessed on any web browser and a smartphone application. The sensor sheet is placed below the mattress and captures data while the user is resting or sleeping and does not require a sensor to be fixed to the body. It consists of the following sub - units: Contactless sensor sheet, Dozee Pod with power cord, 5 V USB Power Adapter, Health data compute server and Web Dashboard/Mobile App. This provides a more comfortable solution for long-term continuous patient monitoring. Continuous monitoring of people's vital signs, in particular Heart Rate (HR) and Respiratory Rate (RR), may provide a mechanism to alert doctors or nurses of clinical deterioration. Monitoring people's vital signs outside an ICU often relies on nursing staff conducting checks at set intervals. The device can reduce the workload for nursing staff in non-ICU wards.

DETAILED DESCRIPTION:
Dozee VS device is intended for the contactless continuous monitoring of vital parameters (Heart Rate and Respiratory Rate), and screening for abnormal changes in these parameters. The device is intended to be used to monitor individuals/patients greater than eighteen (18) years of age (40 kg ≤ weight ≤ 120 kg) and can measure their vital signs during sleep and resting state. The data can be viewed on the dashboard, exported and even be directly transferred to the in-house hospital management software. This protocol aims at verifying the safety and effectiveness of the investigational device in a general-care clinical environment. A similar predicate can be found in the FDA-cleared EarlySense 2.0 (K131379) developed by EarlySense Ltd which shall be used as the predicate device. The device also uses the concept of ballistocardiography and employs piezoelectric sensors to create a contact-less continuous monitoring system which monitors the same vital parameters. It has been sold in over 20 U.S. hospitals since 2013, with no recalls or adverse events reported. According to publicly available clinical results, this system has shown an 86% reduction in Code Blue events, and a 45% reduction in Length of Stay (LoS) in the ICU for patients coming from the medical/surgical unit. The technology employed and the indications for use for the EarlySense device is very similar to the Dozee VS device.

ELIGIBILITY:
Inclusion Criteria:

1. Adults Male or female. (Above 18 years of age)
2. Provide written informed consent.
3. Weight between 40kg/88.18lbs and 120kg/264.55lbs(Above 40 kgs)
4. Are located in a non-ICU hospital setting.
5. Agree to not eat during the testing period (2hours or 10 hours accordingly)

Exclusion Criteria:

1. Are connected to a device which may interfere with the device monitoring in this study.
2. Are receiving any bedside care which may be incompatible with the study procedures.
3. A likely need to receive or undergo a procedure during the testing period.
4. Cannot accept a nasal cannula, or have a monitor lead placed on the chest.
5. Have a significant medical condition in the judgement of the investigator, which may compromise the study testing procedures.
6. Prisoners

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted on 105 subjects in the age group above 18 years regardless of gender. The patients admitted in the hospital will be informed about the study and a written informed consent form will be obtained from them. Dozee will be placed under the mattress of the patient's bed and the data will be collected through the device whenever a patient is on the bed.
  The research team members responsible for data analysis will have access only to the fully anonymised individual-level data and will be blinded to any other patient data, as well as to the components of the calculated scores in the hospital information system.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
RMSD of Investigational Device's Heart Rate and Gold Standard Device's Heart Rate | 12 months
  Record heart rate in the investigational device and patient monitor at the same time every 60 seconds.
  Calculate and compare the root mean square difference (RMSD) per patient and Bland-Alman plot of the heart rate for the investigational device and the gold standard device.
RMSD of Investigational Device's Respiratory Rate and Gold Standard Device's Respiratory Rate | 12 months
  Record respiratory rate in the investigational device and patient monitor at the same time every 60 seconds.
  Calculate and compare the root mean square difference (RMSD) per patient and Bland-Alman plot of the respiratory rate for the investigational device and the gold standard device.
RMSD of Predicate Device's Heart Rate and Gold Standard Device's Heart Rate | 12 months
  Record heart rate in the predicate device and patient monitor at the same time every 60 seconds.
  Calculate and compare the root mean square difference (RMSD) per patient and Bland-Alman plot of the heart rate for the predicate device and the gold standard device.
RMSD of Predicate Device's Respiratory Rate and Gold Standard Device's Respiratory Rate | 12 months
  Record respiratory rate in the investigational device and patient monitor at the same time every 60 seconds.
  Calculate and compare the root mean square difference (RMSD) per patient and Bland-Alman plot of the respiratory rate for the predicate device and the gold standard device.

SECONDARY OUTCOMES:
Motion Notification Accuracy - DUI (%) | 12 months
  Record the time for each instructed movements from manual observation and time for movements notification recorded in the investigational device.
  Calculate the times matched between these two to get the accuracy.
Bed Exit Notification Accuracy - DUI (%) | 12 months
  Record the time for each instructed bed exit from manual observation and time for bed exit notification recorded in the investigational device.
  Calculate the times matched between these two to get the accuracy.
Motion Notification Accuracy - Predicate (%) | 12 months
  Record the time for each instructed movements from manual observation and time for movements notification recorded in the predicate device.
  Calculate the times matched between these two to get the accuracy.
Bed Exit Notification Accuracy - Predicate (%) | 12 months
  Record the time for each instructed bed exit from manual observation and time for bed exit notification recorded in the predicate device.
  Calculate the times matched between these two to get the accuracy.

OTHER OUTCOMES:
Comparison of RMS values of the two primary objectives | 12 months
  Descriptive statistics will be used for capturing study population demographics.
  We will sync timings across the three devices to be able to map concurrent readings and use the longest recorded rate as rate limiting step. (If one device can give 15 second data the oher 30s and the third 60s, we will use 60s as our mark)

CONTACTS AND LOCATIONS:
Locations (1):
- Louisiana State University Health Sciences Center, Shreveport, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
IPD are protected under HIPPA Act of 1996.